CLINICAL TRIAL: NCT01463631
Title: A Phase 1 Study of LY3007113, a p38 MAPK Inhibitor, in Patients With Advanced Cancer
Brief Title: A Study of LY3007113 in Participants With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13513; I5Z-MC-JKBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-10-28; First posted 2011-11-02 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY3007113 (Experimental): Study has a dose escalation phase (Part A) and dose confirmation phase (Part B). Participants in the dose escalation phase will receive 1 of 6 doses of LY3007113 administered orally every 12 hours for at least one cycle. Participants in the dose confirmation phase will receive the maximum tolerated dose from the dose escalation phase administered orally every 12 hours for at least 1 cycle. Three days prior to the start of the first cycle, participants will receive 1 dose at their assigned level to allow for the collection of single dose pharmacokinetics. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criterion is met.
  Interventions: Drug: LY3007113

INTERVENTIONS:
Drug: LY3007113 — Administered orally

SUMMARY:
This study evaluates the safety and tolerability of different doses of an experimental treatment in participants with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological evidence of a diagnosis of cancer that is advanced and/or metastatic for which available standard therapies have failed to provide clinical benefit for their disease
* For Dose Escalation (Part A): cancer, either a solid tumor or a lymphoma
* For Dose Confirmation (Part B): cancer, either a solid tumor or a lymphoma
* Have the presence of measureable or non-measureable disease (Part A) or measureable disease (Part B) as defined by the Response Evaluation Criteria in Solid Tumors or the Revised Response Criteria for Malignant Lymphoma
* Have adequate hematologic, hepatic and renal function
* Have a performance status less than or equal to 2 on the Eastern Cooperative Oncology Group scale
* Have discontinued all previous therapies for cancer (including chemotherapy, radiotherapy, and immunotherapy) for at least 21 days for myelosuppressive agents or 14 days for nonmyelosuppressive agents
* Have an estimated life expectancy of greater than or equal to 12 weeks
* Are able to swallow capsules

Exclusion Criteria:

* Have an echocardiogram with clinically significant abnormalities
* For Dose Escalation (Part A): Have central nervous system malignancy or metastasis
* For Dose Confirmation (Part B): Have symptomatic central nervous system malignancy or metastasis
* Have an acute leukemia
* Have a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and stopped all therapy for that disease for a minimum of 3 years
* Have received an autologous or allogeneic stem-cell transplant within 75 days of the initial dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Monica, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For cohorts 1-3, participants completed the trial if they received at least 75% of planned doses of LY3007113 and completed at least 1 cycle. For Part B, participants completed the trial if they completed at least 2 cycles of study treatment and were assessed for response. (Cycle = 28 days.)
Groups:
- 20 mg LY3007113 (Cohort 1): 20 milligrams (mg) LY3007113 administered orally once every 12 hours on Days 1 through 28. (28-day cycle.) Participants received 2 cycles of treatment. Participants may have received more than 2 cycles of treatment if discontinuation criteria were not met and there was evidence of clinical benefit.
- 40 mg LY3007113 (Cohort 2): 40 mg LY3007113 administered orally once every 12 hours on Days 1 through 28. (28-day cycle.) Participants received 2 cycles of treatment. Participants may have received more than 2 cycles of treatment if discontinuation criteria were not met and there was evidence of clinical benefit.
- 30 mg LY3007113 (Cohort 3); 30 mg LY3007113 (Part B): 30 mg LY3007113 administered orally once every 12 hours on Days 1 through 28. (28-day cycle.) Participants received 2 cycles of treatment. Participants may have received more than 2 cycles of treatment if discontinuation criteria were not met and there was evidence of clinical benefit.
Period: Overall Study
Arm/Group | 20 mg LY3007113 (Cohort 1) | 40 mg LY3007113 (Cohort 2) | 30 mg LY3007113 (Cohort 3) | 30 mg LY3007113 (Part B)
Started | 3 | 4 | 5 | 15
Received at Least One Dose of Study Drug | 3 | 4 | 5 | 15
Completed | 3 | 4 | 4 | 9
Not Completed | 0 | 0 | 1 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug.
Groups:
- 20 mg LY3007113 (Cohort 1): 20 mg LY3007113 administered once orally every 12 hours on Days 1 through 28. (28-day cycle.) Participants may have continued to receive study drug if discontinuation criterion was not met and there was evidence of clinical benefit.
- 40 mg LY3007113 (Cohort 2): 40 mg LY3007113 administered once orally every 12 hours on Days 1 through 28. (28-day cycle.) Participants may have continued to receive study drug if discontinuation criterion was not met and there was evidence of clinical benefit.
- 30 mg LY3007113 (Cohort 3); 30 mg LY3007113 (Part B): 30 mg LY3007113 administered once orally every 12 hours on Days 1 through 28. (28-day cycle.) Participants may have continued to receive study drug if discontinuation criterion was not met and there was evidence of clinical benefit.
- Total: Total of all reporting groups
Arm/Group | 20 mg LY3007113 (Cohort 1) | 40 mg LY3007113 (Cohort 2) | 30 mg LY3007113 (Cohort 3) | 30 mg LY3007113 (Part B) | Total
Number analyzed (Participants) | 3 | 4 | 5 | 15 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4 | 11 | 19
  >=65 years | 1 | 2 | 1 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 8 | 15
  Male | 1 | 1 | 3 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 3 | 3 | 5 | 13 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 2
  White | 2 | 4 | 3 | 13 | 22
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 4 | 5 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Adverse Events (AEs) (Physical Assessments and Clinical Lab Tests)
Description: Data presented are the number of participants who experienced at least one treatment emergent adverse event (TEAE). A TEAE is defined as an event that first occurred or worsened after randomization. A summary of serious AEs and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Event module.
Time Frame: Baseline through Study Completion (up to 170 Days)
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 20 mg LY3007113 (Cohort 1): 20 mg LY3007113 administered orally once every 12 hours on Days 1 through 28. (28-day cycle.) Participants received 2 cycles of treatment. Participants may have received more than 2 cycles of treatment if discontinuation criteria were not met and there was evidence of clinical benefit.
Arm/Group | 20 mg LY3007113 (Cohort 1) | 40 mg LY3007113 (Cohort 2) | 30 mg LY3007113 (Cohort 3) | 30 mg LY3007113 (Part B)
Number analyzed (Participants) | 3 | 4 | 5 | 15
Participants | 2 | 4 | 4 | 8

2. Secondary Outcome: The Percentage of Participants Who Achieved a Best Response of Either Complete Response (CR) or Partial Response (PR): Overall Response Rate (ORR)
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1) criteria. CR was defined as the disappearance of all non-nodal target lesions, with the short axes of any target lymph nodes reduced to <10 millimeters (mm). PR was defined as having at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph nodes), taking as reference the baseline sum diameter without notable worsening of additional tumors that were qualitatively assessed.
Time Frame: Baseline through Study Completion (up to 170 Days)
Population: Participants in Part B who received at least one dose of study drug and were radiologically assessed for tumor response.
Measure: Number; unit: percentage of participants
Arm/Group | 30 mg LY3007113 (Part B)
Number analyzed (Participants) | 13
percentage of participants
  CR | 0
  PR | 0

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-inf]) of Single Dose LY3007113
Time Frame: Cycle 1 Days -3, -2, -1, 1: Predose to 48 hours Postdose
Population: Participants who received at least one dose of study drug and had sufficient evaluable AUC(0-inf) values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Groups:
- 30 mg LY3007113 (Cohort 3 and Part B): 30 mg LY3007113 administered orally once every 12 hours on Days 1 through 28. (28-day cycle.) Participants received 2 cycles of treatment. Participants may have received more than 2 cycles of treatment if discontinuation criteria were not met and there was evidence of clinical benefit.
Arm/Group | 20 mg LY3007113 (Cohort 1) | 40 mg LY3007113 (Cohort 2) | 30 mg LY3007113 (Cohort 3 and Part B)
Number analyzed (Participants) | 3 | 4 | 18
nanogram*hour/milliliter (ng*hr/mL) | 1560 (25) | 2480 (32) | 1810 (67)

4. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From 0 to Tau (AUC[0-tau]) of Multiple Dose LY3007113
Time Frame: Cycle 1 Days 28 and 29, Cycle 2 Day 1: Predose to 24 hours Postdose
Population: Participants who received at least one dose of study drug and had sufficient evaluable AUC(0-tau) values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 20 mg LY3007113 (Cohort 1) | 40 mg LY3007113 (Cohort 2) | 30 mg LY3007113 (Cohort 3 and Part B)
Number analyzed (Participants) | 3 | 4 | 12
ng*hr/mL | 1360 (23) | 3260 (46) | 2070 (68)

5. Secondary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) of LY3007113
Time Frame: Cycle 1 Day -3 (single dose): Predose to 48 hours Postdose; Day 28 (multiple dose): Predose to 24 hours Postdose
Population: Participants who received at least one dose of study drug and had sufficient evaluable Cmax values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 20 mg LY3007113 (Cohort 1) | 40 mg LY3007113 (Cohort 2) | 30 mg LY3007113 (Cohort 3 and Part B)
Number analyzed (Participants) | 3 | 4 | 18
ng/mL
  Single dose | 197 (3) | 296 (66) | 247 (49)
  Multiple dose: number analyzed (Participants) | 3 | 4 | 12
  Multiple dose | 178 (31) | 489 (31) | 386 (64)

ADVERSE EVENTS:
Groups:
- 20 mg LY3007113 (Cohort 1): 20 mg LY3007113 administered orally every 12 hours on Days 1 through 28. (28-day cycle.) Participants may have continued to receive study drug if discontinuation criterion was not met and there was evidence of clinical benefit.
- 40 mg LY3007113 (Cohort 2): 40 mg LY3007113 administered orally every 12 hours on Days 1 through 28. (28-day cycle.) Participants may have continued to receive study drug if discontinuation criterion was not met and there was evidence of clinical benefit.
- 30 mg LY3007113 (Cohort 3); 30 mg LY3007113 (Part B): 30 mg LY3007113 administered orally every 12 hours on Days 1 through 28. (28-day cycle.) Participants may have continued to receive study drug if discontinuation criterion was not met and there was evidence of clinical benefit.
Arm/Group | 20 mg LY3007113 (Cohort 1) | 40 mg LY3007113 (Cohort 2) | 30 mg LY3007113 (Cohort 3) | 30 mg LY3007113 (Part B)
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 2/5 | 5/15
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 5/5 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 mg LY3007113 (Cohort 1) (N=3) | 40 mg LY3007113 (Cohort 2) (N=4) | 30 mg LY3007113 (Cohort 3) (N=5) | 30 mg LY3007113 (Part B) (N=15)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 20 mg LY3007113 (Cohort 1) (N=3) | 40 mg LY3007113 (Cohort 2) (N=4) | 30 mg LY3007113 (Cohort 3) (N=5) | 30 mg LY3007113 (Part B) (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blindness unilateral (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1/7 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (4) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Fatigue (General disorders) | 1 (2) | 2 (2) | 1 (1) | 4 (4)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site rash (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 3 (7) | 1 (1) | 7 (8)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days